CLINICAL TRIAL: NCT06560710
Title: Clinical Characteristics and Surgical Outcomes of Full-thickness Macular Hole Without Focal Vitreomacular Traction.
Status: Completed | Type: Observational
Sponsor: St. Marianna University School of Medicine (Other)
Collaborators: University of Toyama (Other); Takaoka city Hospital (Unknown)
Responsible Party: Principal Investigator, Jiro Kogo, Associate Professor, St. Marianna University School of Medicine
Other Study IDs: MariannaU
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Macular Holes
Keywords: macular hole; epiretinal prolidferation; vitrectomy
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- macular hole without vitreomacular tracation: Vitrectomy
  Interventions: Other: vitrectimy
- Stage 2 macular hole with vitreomacular tracation: Vitrectomy
  Interventions: Other: vitrectimy

INTERVENTIONS:
Other: vitrectimy — Clinical characteristics and surgical outcomes

SUMMARY:
This multicenter, retrospective, observational comparative study. We occasionally encounter FTMHs in which PVD has not been achieved and VMT is absent. These FTMHs cannot be defined by stage in the Gass1) or IVTS3) classification. It is not known whether traction is involved in the development of these atypical macular holes, but they are often classified as Gass stage 2 or 3 according to the size of the hole.

The aim of this study was to investigate the clinical features and surgical outcomes of FTMHs without focal VMT and to discuss possible underlying mechanisms.

DETAILED DESCRIPTION:
The clinical characteristics and surgical outcomes the patients diagnosed with FTMH without focal VMT in the macula (classified as VMT-) are presented, in addition to a comparative analysis of the patients presenting with classic stage 2 FTMH with focal VMT (classified as VMT+) according to international classification criteria.

ELIGIBILITY:
Inclusion Criteria:

- macular hole without posterior vitreous detachment at the fovea

Exclusion Criteria:

* macular hole with posterior vitreous detachment at the fovea
* Stage1.3.4 macular hole
* Macular hole-associated retinal detachment
* Macular hole with subretinal hemorrhage
* Traumatic MH

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
postoperative visual acuity | 1month, 3, 6 and 12 months
  logMAR visual acuity

SECONDARY OUTCOMES:
postoperative status of outer retinal layer in OCT B-scan images | 1month, 3, 6 and 12 months
  External limiting mambrane, Elipsoid zone, Interdegitaion zone

CONTACTS AND LOCATIONS:
Overall Officials: Jiro Kogo, MD PhD, Principal Investigator — Akita University

IPD SHARING:
Plan to Share IPD: No